CLINICAL TRIAL: NCT06707623
Title: Cardiopulmonary Exercise Testing Guided Physiotherapy During Pulmonary Rehabilitation in Patients With Dysfunctional Breathing, a Randomized Controlled Trial
Brief Title: CPET Guided Rehab vs Physiotherapy in Patients With Dysfunctional Breathing
Acronym: DB-REHAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Andreas Asimakos, Consultant Pulmonologist and Director of the Pulmonary Rehabilitation Department, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 564/21-11-24
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Dysfunctional Breathing
Keywords: Dysfunctional Breathing; Pulmonary Rehabilitation; Breathing retraining

STUDY DESIGN:
Intervention Model Description: This is a parallel designed randomized controlled trial with an allocation ratio of 1 control to 1 rehabilitation patient.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): Patients with Dysfunctional Breathing participating in an individualized Rehab Program that will combine exercise and breathing retraining
  Interventions: Other: Pulmonary Rehabilitation
- Physiotherapy Group (Experimental): Patients with dysfunctional breathing in this group will receive respiratory physiotherapy (breathing retraining)
  Interventions: Other: Respiratory Physiotherapy

INTERVENTIONS:
Other: Respiratory Physiotherapy — Physiotherapy will include: Progressive breathing retraining, neurosensory training, nose breathing training, activity modification, inhalation-exhalation ratio training, dynamic respiratory control training and instructions for continuing all of the above training at home. Total 5 sessions in 9 weeks time.
  Arms: Physiotherapy Group
Other: Pulmonary Rehabilitation — Pulmonary Rehabilitation will be completed in 16 sessions (2 times a week for 8 weeks). It will combine exercise with breathing retraining guided by CPET findings regarding erratic breathing pattern and/or hyperventilation.
  Arms: Pulmonary Rehabilitation Group

SUMMARY:
In this study the efficacy of a pulmonary rehabilitation program tailored to the needs of patients with dysfunctional breathing (DB) will be investigated using cardiopulmonary exercise testing. The pulmonary rehabilitation program will be compared with physiotherapy which is currently the mainstream therapy of DB.

DETAILED DESCRIPTION:
Dysfunctional breathing (DB) is a common disorder affecting 9% of the general population and almost 1/3 of patients with underline pulmonary disease such as asthma or COPD. To date physiotherapy utilizing breathing retraining remains the mainstay treatment however, there is lack of evidence regarding the efficacy of these treatments or the superiority of one over the other in terms of symptom relief. Moreover, still there is no consensus on the diagnosis of DB patients and no gold standard diagnostic method exists.

R Boulding et. al. classified DB in to five categories incorporating the main characteristics of patients with DB which are hyperventilation and abnormal/irregular breathing patterns including periodic deep sighing, thoracic dominant breathing, forced abdominal expiration and thoraco-abdominal asynchrony. Patients may demonstrate one or more of the above breathing patterns which are also observed in diseases like asthma, COPD, heart failure, neuromuscular disease and panic/anxiety disorder. To date the main tools for diagnosing/ evaluating DB are expert physiotherapists examination, questionnaires and Cardiopulmonary exercise testing (CPET).

The Nijmegen questionnaire (NQ) has been widely used as a screening tool for DB2 with a cut-off score of ≥23 however, NQ was design for detecting hyperventilation syndrome which is frequent, yet not universal, in DB patients, common in various respiratory conditions and thus poorly agrees with expert respiratory physiotherapists evaluation in detecting DB. The NQ may miss other manifestations of DB like thoracoabdominal asynchrony or apical breathing. The Breathing Pattern Assessment Tool (BPAT) was specifically designed as a semiobjective screening tool for characterization and qualification of the key features of DB namely both hyperventilation and breathing pattern disorders. A cutoff score of ≥4 is highly sensitive (0.92) and specific (0.75) in diagnosing DB9. The Breathing Vigilance (V-Q) Questionnaire was developed to measure breathing vigilance which, if increased, may contribute to DB and could be a therapeutic target. A cut-off score of 16.5 has optimal sensitivity (0.718) and specificity (0.681) in differentiating between high and low DB risk.

CPET could be a valuable tool in diagnosing and assessing dysfunctional breathing. In contrast to questionnaires CPET can be used to objectively assess breathing pattern disorders and provide evidence for further investigations when an underlying disease is suspected. Moreover, as an objective measurement is more reliable in re-assessing DB patients after treatment since there is no "learning effect" from either the patient nor the therapist who both want the therapy to succeed. Assessing end-tidal PCO2 (PETCO2), air blood gases (ABGs) and ventilatory equivalent for VCO2 (VE/VCO2), could help diagnosing DB and ruling out concurrent pathology.

Since breathing retraining remains the main treatment of DB there is an urgent need for further treatment options. Pulmonary rehabilitation has been established as an essential and successful treatment in patients with diseases with high prevalence of DB such as Chronic Obstructive Pulmonary Disease (COPD) and asthma whereas the American Thoracic and European Respiratory Society urge for enhancing the implementation, usage, and Delivery of Pulmonary Rehabilitation in various diseases. We hypothesize that a rehabilitation program with integrated dynamic physiotherapy sessions guided by CPET will be more efficient in the treatment of DB patients than physiotherapy alone. The aim of the present study is to compare a rehabilitation program designed specifically for DB, utilizing CPET for diagnosis and treatment guidance, with breathing retraining alone.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional breathing (DB) diagnosed with CPET.
* Adult patients (>18 years of age)
* Able and willing to attend an outpatient multidisciplinary, supervised rehabilitation program of a total duration of two months (8 weeks).
* Able and willing to attend 5 physiotherapy sessions over a period of 9 weeks.
* Sign an informed consent.

Exclusion Criteria:

* No underling pathology explaining dyspnea and DB in CPET (e.g normal dead space to tidal volume ratio (VD/Vt) and normal alveolar-arterial (A-a) gradient.)
* Patients with COPD
* Patients with uncontrolled asthma
* Patients with post-exertional malaise (PEM).
* Patients that cannot attend an outpatient rehabilitation program like suffering from dementia, chronically paralyzed, with paraplegia, multiple injuries, or other serious orthopaedic problems that cause disability or suffer from very serious underlying diseases such as end-stage cancer, and patients with neurological diseases that cause disability, require specialized rehabilitation clinics and special interventions (speech therapy, kinesiotherapy, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise testing (CPET) | At enrolment and after 8/9 weeks (depends on study arm).

SECONDARY OUTCOMES:
The Nijmegen questionnaire (NQ) | At enrolment and after 8/9 weeks (depends on study arm).
  The Nijmegen questionnaire (NQ) has been widely used as a screening tool for DB with a cut-off score of ≥23 however, NQ was design for detecting hyperventilation syndrome which is frequent, yet not universal, in DB patients. The lowest value is 0 and the highest is 64 with higher scores indicating more severe symptoms and worst outcomes.
The Breathing Pattern Assessment Tool (BPAT) | At enrolment and after 8/9 weeks (depends on study arm).
  The Breathing Pattern Assessment Tool (BPAT) was specifically designed as a semiobjective screening tool for characterization and qualification of the key features of DB namely both hyperventilation and breathing pattern disorders. A cutoff score of ≥4 is highly sensitive (0.92) and specific (0.75) in diagnosing DB. the lowest score is 0 and the highest is 14. Higher scores indicate more symptoms and worst outcomes.
The Breathing Vigilance (V-Q) Questionnaire | At enrolment and after 8/9 weeks (depends on study arm).
  The Breathing Vigilance (V-Q) Questionnaire was developed to measure breathing vigilance which, if increased, may contribute to DB and could be a therapeutic target. A cut-off score of 16.5 has optimal sensitivity (0.718) and specificity (0.681) in differentiating between high and low DB risk . The lowest score is 11 and the highest is 55. Higher scores indicate higher breathing vigilance and worst outcomes.
The Hospital Acquired and Depression Scale (HADS) | At enrolment and after 8/9 weeks (depends on study arm).
  The Hospital Acquired and Depression Scale (HADS) is a 14 items questionnaire that measures anxiety and depression in general medical population. In ARDS survivals the minimal clinically important difference is 2.0-2.5 for the HADS-A and HADS-D. In patients surviving acute lung injury and treated in ICU mean HADS scores remained unchanged in over 2 years follow up (6 for HADS-A and 5 for HADS-D). These values were lower than the threshold of 8 for substantial symptoms of anxiety or depression. The score ranges from 0 to 21 with highest values indicating more anxiety and depression and worst outcomes.
The 36-Item Short Form Health Survey (SF-36) | At enrolment and after 8/9 weeks (depends on study arm).
  The 36-Item Short Form Health Survey (SF-36). The SF-36 is a questionnaire with 36 items that measures health-related quality of life. The 36 questions are separated into 8 scales and 2 composite scales that summarize physical and mental health. The 8 domains are: Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE) and Mental Health (MH). The 2 composites for physical and mental health are Physical Composite Summary (PCS) and Mental Composite Summary (MCS). Domain and summary components scores range from 0 to 100, with higher score represents better quality of life and well - being. With scoring algorithms, score from all the domains place on scales with mean scores equal to 50.
Modified Medical Research Council (mMRC) Dyspnea Scale | At enrolment and after 8/9 weeks (depends on study arm).
  The Modified Medical Research Council (mMRC) Dyspnea Scale is a 5 point scale based on the sensation of dyspnea during patients daily activities with 0 identifying patients that only get breathless with strenuous exercise and 4 patients that are too breathless to get dressed or leave home. MMRC scale is mostly used to stratify patients based on symptoms and due το limited levels of classification is frequently unable to detect small changes, yet both groups in the present study showed statistically significant changes.
Airway occlusion pressure P0.1 | At enrolment and after 8/9 weeks (depends on study arm).
  Airway occlusion pressure (P0.1) is the drop in airway pressure (Paw) 100 milliseconds after the onset of inspiration during an end-expiratory occlusion of the airway. It is, in theory, a reliable measure of respiratory drive because the brevity of the occlusion explains that it is not affected by patient's response to the occlusion and it is independent of respiratory mechanics.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary Rehabilitation Unit, 1st Department of Critical Care and Pulmonary Services Evangelismos Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data is prohibited by the hospital's patient privacy policy. Patient data may only be used for the purposes of this study.

REFERENCES:
- [Background] van Dixhoorn J, Duivenvoorden HJ. Efficacy of Nijmegen Questionnaire in recognition of the hyperventilation syndrome. J Psychosom Res. 1985;29(2):199-206. doi: 10.1016/0022-3999(85)90042-x. PMID 4009520
- [Background] Todd S, Walsted ES, Grillo L, Livingston R, Menzies-Gow A, Hull JH. Novel assessment tool to detect breathing pattern disorder in patients with refractory asthma. Respirology. 2018 Mar;23(3):284-290. doi: 10.1111/resp.13173. Epub 2017 Sep 14. PMID 28905471
- [Background] Steinmann J, Lewis A, Ellmers TJ, Jones M, MacBean V, Kal E. Validating the Breathing Vigilance Questionnaire for use in dysfunctional breathing. Eur Respir J. 2023 Jun 8;61(6):2300031. doi: 10.1183/13993003.00031-2023. Print 2023 Jun. PMID 37024133
- [Background] Genecand L, Altarelli M, Binkova A, Loew S, Vaudan S, Gex G, Bridevaux PO, Fresard I. Dysfunctional breathing symptoms, functional impact and quality of life in patients with long COVID-19: a prospective case series. BMJ Open Respir Res. 2023 Jul;10(1):e001770. doi: 10.1136/bmjresp-2023-001770. PMID 37433720